CLINICAL TRIAL: NCT00608881
Title: Coenzyme Q10 in Huntington's Disease (HD)
Acronym: 2CARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility analysis failed to showed likelihoo of benefit of CoQ 2400 mg/day.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of Rochester (Other)
Responsible Party: Principal Investigator, Merit E. Cudkowicz, MD, Julieanne Dorn Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2CARE 01.00; 5U01NS052592 (NIH); 5R01NS052619 (NIH)
Record Dates: First submitted 2008-02-04; First posted 2008-02-06 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease; Huntington disease; HD; coenzyme Q10; CoQ
MeSH Terms: conditions — Huntington Disease | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - coenzyme Q10 2400 mg/day (Active Comparator): Randomized to active treatment (coenzyme Q10 2400 mg/day)
  Interventions: Drug: coenzyme Q10
- B - Placebo (Placebo Comparator): Randomized to placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: coenzyme Q10 — 4 - 300 mg CoQ chewable wafers taken orally twice a day
  Other Names: CoQ
  Arms: A - coenzyme Q10 2400 mg/day
Other: placebo — an inactive substance
  Arms: B - Placebo

SUMMARY:
The goals of this trial are to determine if coenzyme Q10 is effective in slowing the worsening symptoms of Huntington's disease and to learn about the safety and acceptability of long-term coenzyme Q10 use by determining its effects on people with Huntington's disease.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a slowly progressive disorder that devastates the lives of those affected and their families. There are no treatments that slow the progression of HD, only mildly effective symptomatic therapies are available.

The purpose of this trial is to find out if coenzyme Q10 (CoQ) is effective in slowing the worsening symptoms of HD. In this study, researchers also will learn about the safety and acceptability of long-term CoQ use by determining its effects on people with HD.

Participants in this trial will be randomly chosen to one of two groups. Group 1 will receive CoQ (2400 mg/day), and group 2 will receive a placebo (an inactive substance). Researchers will compare the change in total functional capacity (TFC)-a measure of functional disability-in the two groups. The TFC is a valid and reliable measure of disease progression and is particularly responsive to change in the early and mid-stages of HD. Researchers will also compare the changes in other components of the Unified Huntington's Disease Rating Scale '99 (UHDRS) including: the total motor score, total behavioral frequency score, total behavior frequency X severity score, verbal fluency test, symbol digit modalities test, Stroop, interference test, functional checklist, and independence scale scores. The groups will also be compared with respect to tolerability, adverse events, vital signs, and laboratory test results as measures of safety.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment into this study, subjects must meet the following eligibility criteria within 28 days prior to randomization:

* Subjects must have clinical features of HD and a confirmed family history of HD, OR a CAG repeat expansion ≥ 36.
* TFC > 9.
* Must be ambulatory and not require skilled nursing care.
* Age ≥ 16 years.
* Women must not be able to become pregnant (e.g., post menopausal, surgically sterile or using adequate birth control methods for the duration of the study).
* If psychotropic medications are taken (e.g., anxiolytics, hypnotics, benzodiazepines, antidepressants), they must be at a stable dosage for four weeks prior to randomization and should be maintained at a constant dosage throughout the study, as possible. (Note: stable dosing of tetrabenazine is allowable.) Any changes to these medications mandated by clinical conditions will be systematically recorded and the subject will be permitted to remain in the trial.
* Able to give informed consent and comply with trial procedures
* Able to take oral medication.
* May be required to identify an informant or caregiver who will be willing and able to supervise the daily dosing of study medications and to maintain control of study medications in the home.
* A designated individual will be identified by the subject to participate in the ongoing consent process should the subject's cognitive capacity to consent become compromised during participation in the study.

Exclusion Criteria:

* History or known sensitivity of intolerability to CoQ.
* Exposure to any investigational drug within 30 days of the Baseline visit.
* Clinical evidence of unstable medical illness in the investigator's judgment.
* Unstable psychiatric illness defined as psychosis (hallucinations or delusions), untreated major depression or suicidal ideation within 90 days of the Baseline visit.
* Substance (alcohol or drug) abuse within one year of the Baseline visit.
* Women who are pregnant or breastfeeding.
* Use of supplemental coenzyme Q10 within 30 days prior to the Baseline visit
* Clinically serious abnormalities in the screening laboratory studies (Screening creatinine greater than 2.0, alanine aminotransferase (ALT) or total bilirubin greater than 3 times the upper limit of normal, absolute neutrophil count of ≤1000/ul, platelet concentration of <100,000/ul, hematocrit level of <33 for female or <35 for male, or coagulation tests > 1.5 time upper limit of normal).
* Known allergy to FD&C yellow #5 or any other ingredient in the study drug (active and placebo)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2008-03; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD MSc, Principal Investigator — Massachusetts General Hospital; Michael McDermott, PhD, Principal Investigator — University of Rochester, Biostatistics; Karl Kieburtz, MD MPH, Principal Investigator — Director, Clinical Trials Coordination Center, University of Rochester
Locations (49):
- United States (41):
  - University of Alabama At Birmingham, Pediatric Neurology Childrens, Harbor Bldg Suite 314, 1600 7Th Avenue South, Birmingham, Alabama
  - Mayo Clinic Arizona, 13400 East Shea Boulevard, Csu-Cp21B, Scottsdale, Arizona
  - WASHINGTON REGIONAL MEDICAL CENTER, 3215 N. North Hills Blvd, Fayetteville, Arkansas
  - University of California Irvine, Department of Neurology, 100 Irvine Hall, Irvine, California
  - University of California Davis, Medical Center Dept of Neurology, Acc Building Suite 3700, 4860 Y Street, Sacramento, California
  - Colorado Neurological Institute, Movement Disorders Center, 701 East Hampden Avenue Suite 510, Littleton, Colorado
  - University of Florida Center for Movement Disorders and Neurorestoration, 3450 Hull Road, 4th Floor, Gainesville, Florida
  - UNIVERSITY OF MIAMI, 1150 NW 14th STREET, #401, Miami, Florida
  - University of South Florida, College of Medicine Dept of Neurology, 12901 Bruce B Downs Blvd Mdc-55, Tampa, Florida
  - Emory University, Wesley Woods Center, 1841 Clifton Road NE Room 314, Atlanta, Georgia
  - Idaho Elks Rehabilitation Hospital, 600 North Robbins Road, Boise, Idaho
  - Rush University Medical Center, Department of Neurological Sciences, 1725 West Harrison Suite 755, Chicago, Illinois
  - Indiana University School of Medicine, Outpatient Clinical Research Facility, 535 Barnhill Drive Room #150, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, 200 Hawkins Road, Room W263 General Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Department of Neurology, 3599 Rainbow Blvd Mail Stop 2012, Kansas City, Kansas
  - Hereditary Neurological Disease Centre (Hndc),3223 N. Webb, Suite 4, Wichita, Kansas
  - University of Maryland School of Medicine, 22 South Greene Street, N4 W49-B, Baltimore, Maryland
  - Johns Hopkins University, 600 North Wolfe Street, Meyer 2-181, Baltimore, Maryland
  - Boston University School of Medicine, Department of Neurology, 715 Albany Street C329, Boston, Massachusetts
  - Massachusetts General Hospital, 149 13Th Street Suite 2241, Charlestown, Massachusetts
  - University of Michigan, 1500 E Medical Center Drive, B1 H202 Nuclear Medicine, Ann Arbor, Michigan
  - Struthers Parkinson'S Center, 6701 Country Club Drive, Golden Valley, Minnesota
  - Washington University School of Medicine, Box 8111, 660 South Euclid, St Louis, Missouri
  - University of Las Vegas School of Medicine, 1707 W. Charleston Blvd, Suite 220, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Nj Neuroscience Institute, Jfk Medical Center, 65 James Street, Edison, New Jersey
  - Albany Medical College, Parkinson'S Disease & Movement Disorders Ctr, Albany, New York
  - North Shore-Lij Health System, 350 Community Drive Room 110, Research Institute, Manhasset, New York
  - Columbia University, Sergievsky Center P&S Box 16, 630 West 168Th Street, New York, New York
  - University of Rochester, Department of Neurology, 919 Westfall Road Building C Suite 220, Rochester, New York
  - Duke University, 932 Morreene Road #213, Durham, North Carolina
  - Wake Forest University, Baptist Med Center, Department of Neurology, Medical Center Boulevard, Winston-Salem, North Carolina
  - University of Cincinnati/Cincinnati Children'S Hospital, 222 Piedmont Avenue, Suite 3200, Cincinnati, Ohio
  - OHIO STATE UNIVERSITY , 2006 Kenny Road, Columbus, Ohio
  - ST. LUKE'S HOSPITAL, 240 Centronia Road, Allentown, Pennsylvania
  - University of Pennsylvania, Pennsylvania Hospital Department of Neurology , 330 South 9Th Street, Philadelphia, Pennsylvania
  - University of Pittsburgh Kaufmann Medical Building, 3471 Fifth Avunue, Suite 811, Pittsburgh, Pennsylvania
  - BUTLER HOSPTIAL MOVEMENT DISORDER PROGRAM, 345 Blackstone Boulevard, Providence, Rhode Island
  - The University of Tennesee Health Science Cen, 855 Monroe Avenue, Department of Neurology, Room 415 Link Bldg, Memphis, Tennessee
  - UN oF TEXAS SOUTHWESTERN MED CENTER DALLAS, 5323 HARRY HINES BOULEVARD H1.108, Dallas, Texas
  - Baylor College of Medicine, 6550 Fannin Suite 1801, Houston, Texas
- Westmead Hospital, Department of Neurology Level 1, Po Box 533, Wentworthville, New South Wales, Australia
- Canada (7):
  - University of Calgary, Heritage Medical Research Clinic, Trw Bldg 5 Floor, 3280 Hospital Dri. NW, Calgary, Alberta
  - University of Alberta, Glenrose Rehab Hosp, Movement Disorder Clinic , Rm 0601 Gleneast 10230 - 111 Avenue, Edmonton, Alberta
  - Department of Medical Genetics, Ubc Hospital, Room S179-2211 Westbrook Mall, Vancouver, British Columbia
  - London Health Sciences Centre, University Hospital, 339 Windermere Road, London, Ontario
  - Centre For Movement Disorders, 2780 Bur Oak Avenue, Markham, Ontario
  - NORTH YORK GENERAL HOSPITAL (2), 4001 Leslie Street, Toronto, Ontario
  - North York General Hospital, 4001 Leslie Street, Toronto, Ontario

REFERENCES:
- [Background] Kowall N, Ferrante R, Martin J. Patterns of cell loss in Huntington's disease. Trends in Neurosciences 1987;10:24-29.
- [Background] Riley D, Lang A. Movement Disorders. In: Bradley W, Daroff R, Fenichel G, eds. Neurology in Clinical Practice. The Neurological Disorders. Boston: Butterworth-Heinemann, 1991: 1563-1601.
- [Background] Adams P, Falek A, Arnold J. Huntington disease in Georgia: age at onset. Am J Hum Genet. 1988 Nov;43(5):695-704. PMID 2973230
- [Background] Conneally PM. Huntington disease: genetics and epidemiology. Am J Hum Genet. 1984 May;36(3):506-26. PMID 6233902
- [Background] Harper PS. The epidemiology of Huntington's disease. Hum Genet. 1992 Jun;89(4):365-76. doi: 10.1007/BF00194305. PMID 1535611
- [Background] Tanner CM, Goldman SM. Epidemiology of movement disorders. Curr Opin Neurol. 1994 Aug;7(4):340-5. doi: 10.1097/00019052-199408000-00011. No abstract available. PMID 7952243
- [Background] Young AB, Shoulson I, Penney JB, Starosta-Rubinstein S, Gomez F, Travers H, Ramos-Arroyo MA, Snodgrass SR, Bonilla E, Moreno H, et al. Huntington's disease in Venezuela: neurologic features and functional decline. Neurology. 1986 Feb;36(2):244-9. doi: 10.1212/wnl.36.2.244. PMID 2935747
- [Background] Bruyn G. Huntington's chorea: Historical clinical and laboratory synopsis. In: Vinken P, Bruyn G, eds. Handbook of Clinical Neurology. Amsterdam, 1968: 298-378.
- [Background] Leigh RJ, Newman SA, Folstein SE, Lasker AG, Jensen BA. Abnormal ocular motor control in Huntington's disease. Neurology. 1983 Oct;33(10):1268-75. doi: 10.1212/wnl.33.10.1268. PMID 6225033
- [Background] Caine ED, Hunt RD, Weingartner H, Ebert MH. Huntington's dementia. Clinical and neuropsychological features. Arch Gen Psychiatry. 1978 Mar;35(3):377-84. doi: 10.1001/archpsyc.1978.01770270127013. PMID 153122
- [Background] Bamford KA, Caine ED, Kido DK, Plassche WM, Shoulson I. Clinical-pathologic correlation in Huntington's disease: a neuropsychological and computed tomography study. Neurology. 1989 Jun;39(6):796-801. doi: 10.1212/wnl.39.6.796. PMID 2524678
- [Background] Sorensen SA, Fenger K. Causes of death in patients with Huntington's disease and in unaffected first degree relatives. J Med Genet. 1992 Dec;29(12):911-4. doi: 10.1136/jmg.29.12.911. PMID 1479606
- [Background] Oliver JE. Huntington's chorea in Northamptonshire. Br J Psychiatry. 1970 Mar;116(532):241-53. doi: 10.1192/bjp.116.532.241. No abstract available. PMID 4244787
- [Background] Greenamyre J, Shoulson I. Huntington's Disease. In: Calne D, ed. Neurodegenerative Diseases. Philadelphia: WB Saunders, 1994: 685-704.
- [Background] Shoulson I, Fahn S. Huntington disease: clinical care and evaluation. Neurology. 1979 Jan;29(1):1-3. doi: 10.1212/wnl.29.1.1. No abstract available. PMID 154626
- [Background] Feigin A, Kieburtz K, Bordwell K, Como P, Steinberg K, Sotack J, Zimmerman C, Hickey C, Orme C, Shoulson I. Functional decline in Huntington's disease. Mov Disord. 1995 Mar;10(2):211-4. doi: 10.1002/mds.870100213. PMID 7753064
- [Background] Myers RH, Sax DS, Koroshetz WJ, Mastromauro C, Cupples LA, Kiely DK, Pettengill FK, Bird ED. Factors associated with slow progression in Huntington's disease. Arch Neurol. 1991 Aug;48(8):800-4. doi: 10.1001/archneur.1991.00530200036015. PMID 1832854
- [Background] Penney JB Jr, Young AB, Shoulson I, Starosta-Rubenstein S, Snodgrass SR, Sanchez-Ramos J, Ramos-Arroyo M, Gomez F, Penchaszadeh G, Alvir J, et al. Huntington's disease in Venezuela: 7 years of follow-up on symptomatic and asymptomatic individuals. Mov Disord. 1990;5(2):93-9. doi: 10.1002/mds.870050202. PMID 2139171
- [Background] Young AB, Penney JB, Starosta-Rubinstein S, Markel DS, Berent S, Giordani B, Ehrenkaufer R, Jewett D, Hichwa R. PET scan investigations of Huntington's disease: cerebral metabolic correlates of neurological features and functional decline. Ann Neurol. 1986 Sep;20(3):296-303. doi: 10.1002/ana.410200305. PMID 2945510
- [Background] Kido D, Shoulson I, Manzione J, Harnish P. Measurement of caudate nucleus and putamen atrophy in patients with Huntington's disease. Neuroradiology 1991;33:604-606.
- [Background] Mazziotta JC. Huntington's disease: studies with structural imaging techniques and positron emission tomography. Semin Neurol. 1989 Dec;9(4):360-9. doi: 10.1055/s-2008-1041346. No abstract available. PMID 2534934
- [Background] Beal MF, Ferrante RJ. Experimental therapeutics in transgenic mouse models of Huntington's disease. Nat Rev Neurosci. 2004 May;5(5):373-84. doi: 10.1038/nrn1386. No abstract available. PMID 15100720
- [Background] A novel gene containing a trinucleotide repeat that is expanded and unstable on Huntington's disease chromosomes. The Huntington's Disease Collaborative Research Group. Cell. 1993 Mar 26;72(6):971-83. doi: 10.1016/0092-8674(93)90585-e. PMID 8458085
- [Background] Tabrizi SJ, Workman J, Hart PE, Mangiarini L, Mahal A, Bates G, Cooper JM, Schapira AH. Mitochondrial dysfunction and free radical damage in the Huntington R6/2 transgenic mouse. Ann Neurol. 2000 Jan;47(1):80-6. doi: 10.1002/1531-8249(200001)47:13.3.co;2-b. PMID 10632104
- [Background] Cha JH. Transcriptional dysregulation in Huntington's disease. Trends Neurosci. 2000 Sep;23(9):387-92. doi: 10.1016/s0166-2236(00)01609-x. PMID 10941183
- [Background] Ona VO, Li M, Vonsattel JP, Andrews LJ, Khan SQ, Chung WM, Frey AS, Menon AS, Li XJ, Stieg PE, Yuan J, Penney JB, Young AB, Cha JH, Friedlander RM. Inhibition of caspase-1 slows disease progression in a mouse model of Huntington's disease. Nature. 1999 May 20;399(6733):263-7. doi: 10.1038/20446. PMID 10353249
- [Background] Chen M, Ona VO, Li M, Ferrante RJ, Fink KB, Zhu S, Bian J, Guo L, Farrell LA, Hersch SM, Hobbs W, Vonsattel JP, Cha JH, Friedlander RM. Minocycline inhibits caspase-1 and caspase-3 expression and delays mortality in a transgenic mouse model of Huntington disease. Nat Med. 2000 Jul;6(7):797-801. doi: 10.1038/77528. PMID 10888929
- [Background] Beal MF, Hyman BT, Koroshetz W. Do defects in mitochondrial energy metabolism underlie the pathology of neurodegenerative diseases? Trends Neurosci. 1993 Apr;16(4):125-31. doi: 10.1016/0166-2236(93)90117-5. PMID 7682343
- [Background] Wellington CL, Ellerby LM, Hackam AS, Margolis RL, Trifiro MA, Singaraja R, McCutcheon K, Salvesen GS, Propp SS, Bromm M, Rowland KJ, Zhang T, Rasper D, Roy S, Thornberry N, Pinsky L, Kakizuka A, Ross CA, Nicholson DW, Bredesen DE, Hayden MR. Caspase cleavage of gene products associated with triplet expansion disorders generates truncated fragments containing the polyglutamine tract. J Biol Chem. 1998 Apr 10;273(15):9158-67. doi: 10.1074/jbc.273.15.9158. PMID 9535906
- [Background] Brouillet E, Hantraye P, Ferrante RJ, Dolan R, Leroy-Willig A, Kowall NW, Beal MF. Chronic mitochondrial energy impairment produces selective striatal degeneration and abnormal choreiform movements in primates. Proc Natl Acad Sci U S A. 1995 Jul 18;92(15):7105-9. doi: 10.1073/pnas.92.15.7105. PMID 7624378
- [Background] Gu M, Gash MT, Mann VM, Javoy-Agid F, Cooper JM, Schapira AH. Mitochondrial defect in Huntington's disease caudate nucleus. Ann Neurol. 1996 Mar;39(3):385-9. doi: 10.1002/ana.410390317. PMID 8602759
- [Background] Koroshetz WJ, Jenkins BG, Rosen BR, Beal MF. Energy metabolism defects in Huntington's disease and effects of coenzyme Q10. Ann Neurol. 1997 Feb;41(2):160-5. doi: 10.1002/ana.410410206. PMID 9029064
- [Background] Sawa A, Wiegand GW, Cooper J, Margolis RL, Sharp AH, Lawler JF Jr, Greenamyre JT, Snyder SH, Ross CA. Increased apoptosis of Huntington disease lymphoblasts associated with repeat length-dependent mitochondrial depolarization. Nat Med. 1999 Oct;5(10):1194-8. doi: 10.1038/13518. PMID 10502825
- [Background] Jenkins BG, Koroshetz WJ, Beal MF, Rosen BR. Evidence for impairment of energy metabolism in vivo in Huntington's disease using localized 1H NMR spectroscopy. Neurology. 1993 Dec;43(12):2689-95. doi: 10.1212/wnl.43.12.2689. PMID 8255479
- [Background] Lodi R, Schapira AH, Manners D, Styles P, Wood NW, Taylor DJ, Warner TT. Abnormal in vivo skeletal muscle energy metabolism in Huntington's disease and dentatorubropallidoluysian atrophy. Ann Neurol. 2000 Jul;48(1):72-6. PMID 10894218
- [Background] Panov AV, Gutekunst CA, Leavitt BR, Hayden MR, Burke JR, Strittmatter WJ, Greenamyre JT. Early mitochondrial calcium defects in Huntington's disease are a direct effect of polyglutamines. Nat Neurosci. 2002 Aug;5(8):731-6. doi: 10.1038/nn884. PMID 12089530
- [Background] Gines S, Seong IS, Fossale E, Ivanova E, Trettel F, Gusella JF, Wheeler VC, Persichetti F, MacDonald ME. Specific progressive cAMP reduction implicates energy deficit in presymptomatic Huntington's disease knock-in mice. Hum Mol Genet. 2003 Mar 1;12(5):497-508. doi: 10.1093/hmg/ddg046. PMID 12588797
- [Background] Browne SE, Bowling AC, MacGarvey U, Baik MJ, Berger SC, Muqit MM, Bird ED, Beal MF. Oxidative damage and metabolic dysfunction in Huntington's disease: selective vulnerability of the basal ganglia. Ann Neurol. 1997 May;41(5):646-53. doi: 10.1002/ana.410410514. PMID 9153527
- [Background] Ferrante RJ, Andreassen OA, Jenkins BG, Dedeoglu A, Kuemmerle S, Kubilus JK, Kaddurah-Daouk R, Hersch SM, Beal MF. Neuroprotective effects of creatine in a transgenic mouse model of Huntington's disease. J Neurosci. 2000 Jun 15;20(12):4389-97. doi: 10.1523/JNEUROSCI.20-12-04389.2000. PMID 10844007
- [Background] Ferrante RJ, Andreassen OA, Dedeoglu A, Ferrante KL, Jenkins BG, Hersch SM, Beal MF. Therapeutic effects of coenzyme Q10 and remacemide in transgenic mouse models of Huntington's disease. J Neurosci. 2002 Mar 1;22(5):1592-9. doi: 10.1523/JNEUROSCI.22-05-01592.2002. PMID 11880489
- [Background] Dedeoglu A, Kubilus JK, Yang L, Ferrante KL, Hersch SM, Beal MF, Ferrante RJ. Creatine therapy provides neuroprotection after onset of clinical symptoms in Huntington's disease transgenic mice. J Neurochem. 2003 Jun;85(6):1359-67. doi: 10.1046/j.1471-4159.2003.01706.x. PMID 12787055
- [Background] Schilling G, Coonfield ML, Ross CA, Borchelt DR. Coenzyme Q10 and remacemide hydrochloride ameliorate motor deficits in a Huntington's disease transgenic mouse model. Neurosci Lett. 2001 Nov 27;315(3):149-53. doi: 10.1016/s0304-3940(01)02326-6. PMID 11716985
- [Background] Matthews RT, Yang L, Browne S, Baik M, Beal MF. Coenzyme Q10 administration increases brain mitochondrial concentrations and exerts neuroprotective effects. Proc Natl Acad Sci U S A. 1998 Jul 21;95(15):8892-7. doi: 10.1073/pnas.95.15.8892. PMID 9671775
- [Background] Beal MF, Henshaw DR, Jenkins BG, Rosen BR, Schulz JB. Coenzyme Q10 and nicotinamide block striatal lesions produced by the mitochondrial toxin malonate. Ann Neurol. 1994 Dec;36(6):882-8. doi: 10.1002/ana.410360613. PMID 7998775
- [Background] Pepping J. Coenzyme Q10. Am J Health Syst Pharm. 1999 Mar 15;56(6):519-21. doi: 10.1093/ajhp/56.6.519. No abstract available. PMID 10192685
- [Background] Musumeci O, Naini A, Slonim AE, Skavin N, Hadjigeorgiou GL, Krawiecki N, Weissman BM, Tsao CY, Mendell JR, Shanske S, De Vivo DC, Hirano M, DiMauro S. Familial cerebellar ataxia with muscle coenzyme Q10 deficiency. Neurology. 2001 Apr 10;56(7):849-55. doi: 10.1212/wnl.56.7.849. PMID 11294920
- [Background] Ernster L, Dallner G. Biochemical, physiological and medical aspects of ubiquinone function. Biochim Biophys Acta. 1995 May 24;1271(1):195-204. doi: 10.1016/0925-4439(95)00028-3. PMID 7599208
- [Background] Yamagami T, Okishio T, Toyama S, Kishi T. Correlation of serum coenzyme Q10 level and leukocute complex II activity in nformal and cardiovascular patients. In: Folkers K, Yamagami T, eds. Biomedical and clinical aspects of coenzyme Q: Elsevier Science Publishers, 1981: 79-89.
- [Background] Soderberg M, Edlund C, Kristensson K, Dallner G. Lipid compositions of different regions of the human brain during aging. J Neurochem. 1990 Feb;54(2):415-23. doi: 10.1111/j.1471-4159.1990.tb01889.x. PMID 2299344
- [Background] Peyser CE, Folstein M, Chase GA, Starkstein S, Brandt J, Cockrell JR, Bylsma F, Coyle JT, McHugh PR, Folstein SE. Trial of d-alpha-tocopherol in Huntington's disease. Am J Psychiatry. 1995 Dec;152(12):1771-5. doi: 10.1176/ajp.152.12.1771. PMID 8526244
- [Background] Ranen NG, Peyser CE, Coyle JT, Bylsma FW, Sherr M, Day L, Folstein MF, Brandt J, Ross CA, Folstein SE. A controlled trial of idebenone in Huntington's disease. Mov Disord. 1996 Sep;11(5):549-54. doi: 10.1002/mds.870110510. PMID 8866496
- [Background] Kremer B, Clark CM, Almqvist EW, Raymond LA, Graf P, Jacova C, Mezei M, Hardy MA, Snow B, Martin W, Hayden MR. Influence of lamotrigine on progression of early Huntington disease: a randomized clinical trial. Neurology. 1999 Sep 22;53(5):1000-11. doi: 10.1212/wnl.53.5.1000. PMID 10496259
- [Background] Puri BK, Leavitt BR, Hayden MR, Ross CA, Rosenblatt A, Greenamyre JT, Hersch S, Vaddadi KS, Sword A, Horrobin DF, Manku M, Murck H. Ethyl-EPA in Huntington disease: a double-blind, randomized, placebo-controlled trial. Neurology. 2005 Jul 26;65(2):286-92. doi: 10.1212/01.wnl.0000169025.09670.6d. PMID 16043801
- [Background] Dubois B, Brand M, Garcia de Yebenes J, et al. European-Huntington's-disease-Initiative (EHDI)-Trial: Objectives, design, and description of the study population at the end of inclusion. Mov Dis 2002;17:S319.
- [Background] Bogentoft C, Edelund P, Olsson B, Widlund L, Westensen K. Biopharmaceutical aspects of intraveneous and oral administration of coenzyme Q10. In: Folkers K, Littarru G, Yamagami T, eds. Biomedical and clinical aspects of coenzyme Q.: Elsevier Science Publishers, 1991: 215-224.
- [Background] Lucker P, Wetselsberg N, Hennings G, Rehn D. Pharmacokinetics of coenzyme ubidecarenone in healthy volunteers. In: Folkers K, Littarru G, Yamagami T, eds. Biomedical and clinical aspects of coenzyme Q: Elsevier Science Publishers, 1984: 143-151.
- [Background] Mohr D, Bowry VW, Stocker R. Dietary supplementation with coenzyme Q10 results in increased levels of ubiquinol-10 within circulating lipoproteins and increased resistance of human low-density lipoprotein to the initiation of lipid peroxidation. Biochim Biophys Acta. 1992 Jun 26;1126(3):247-54. doi: 10.1016/0005-2760(92)90237-p. PMID 1637852
- [Background] Micromedex. Ubidecarenone drug monograph. Engelwood 1995 May; Update 1998 Mar.
- [Background] Zhang Y, Aberg F, Appelkvist EL, Dallner G, Ernster L. Uptake of dietary coenzyme Q supplement is limited in rats. J Nutr. 1995 Mar;125(3):446-53. doi: 10.1093/jn/125.3.446. PMID 7876919
- [Background] Weber C. Dietary intake and absorption of coenzyme Q. In: Kagan V, Quinn P, eds. Coenzyme Q: Molecular Mechanisms in Health and Disease. Boca Raton: CRC Press, 2001:209-215.
- [Background] Rundek T, Naini A, Sacco R, Coates K, DiMauro S. Atorvastatin decreases the coenzyme Q10 level in the blood of patients at risk for cardiovascular disease and stroke. Arch Neurol. 2004 Jun;61(6):889-92. doi: 10.1001/archneur.61.6.889. PMID 15210526
- [Background] Saito Y, Kubo H, Bujo H, Yamamoto Y. The changes in plasma coenzyme Q10 level during the statin therapy for hypercholesterolemic patients. In: Second Conference of the International Coenzyme Q10 Association.; 2000, 2000: 59.
- [Background] De Pinieux G, Chariot P, Ammi-Said M, Louarn F, Lejonc JL, Astier A, Jacotot B, Gherardi R. Lipid-lowering drugs and mitochondrial function: effects of HMG-CoA reductase inhibitors on serum ubiquinone and blood lactate/pyruvate ratio. Br J Clin Pharmacol. 1996 Sep;42(3):333-7. doi: 10.1046/j.1365-2125.1996.04178.x. PMID 8877024
- [Background] Watts GF, Castelluccio C, Rice-Evans C, Taub NA, Baum H, Quinn PJ. Plasma coenzyme Q (ubiquinone) concentrations in patients treated with simvastatin. J Clin Pathol. 1993 Nov;46(11):1055-7. doi: 10.1136/jcp.46.11.1055. PMID 8254097
- [Background] Laaksonen R, Jokelainen K, Laakso J, Sahi T, Harkonen M, Tikkanen MJ, Himberg JJ. The effect of simvastatin treatment on natural antioxidants in low-density lipoproteins and high-energy phosphates and ubiquinone in skeletal muscle. Am J Cardiol. 1996 Apr 15;77(10):851-4. doi: 10.1016/S0002-9149(97)89180-1. PMID 8623738
- [Background] Huntington Study Group. Minocycline safety and tolerability in Huntington disease. Neurology. 2004 Aug 10;63(3):547-9. doi: 10.1212/01.wnl.0000133403.30559.ff. PMID 15304592
- [Background] Langsjoen H, Langsjoen P, Langsjoen P, Willis R, Folkers K. Usefulness of coenzyme Q10 in clinical cardiology: a long-term study. Mol Aspects Med. 1994;15 Suppl:s165-75. doi: 10.1016/0098-2997(94)90026-4. PMID 7752828
- [Background] Ogasahara S, Engel AG, Frens D, Mack D. Muscle coenzyme Q deficiency in familial mitochondrial encephalomyopathy. Proc Natl Acad Sci U S A. 1989 Apr;86(7):2379-82. doi: 10.1073/pnas.86.7.2379. PMID 2928337
- [Background] Di Giovanni S, Mirabella M, Spinazzola A, Crociani P, Silvestri G, Broccolini A, Tonali P, Di Mauro S, Servidei S. Coenzyme Q10 reverses pathological phenotype and reduces apoptosis in familial CoQ10 deficiency. Neurology. 2001 Aug 14;57(3):515-8. doi: 10.1212/wnl.57.3.515. PMID 11502923
- [Background] Lodi R, Hart PE, Rajagopalan B, Taylor DJ, Crilley JG, Bradley JL, Blamire AM, Manners D, Styles P, Schapira AH, Cooper JM. Antioxidant treatment improves in vivo cardiac and skeletal muscle bioenergetics in patients with Friedreich's ataxia. Ann Neurol. 2001 May;49(5):590-6. PMID 11357949
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Shults CW, Flint Beal M, Song D, Fontaine D. Pilot trial of high dosages of coenzyme Q10 in patients with Parkinson's disease. Exp Neurol. 2004 Aug;188(2):491-4. doi: 10.1016/j.expneurol.2004.05.003. PMID 15246848
- [Background] Greenberg S, Frishman WH. Co-enzyme Q10: a new drug for cardiovascular disease. J Clin Pharmacol. 1990 Jul;30(7):596-608. doi: 10.1002/j.1552-4604.1990.tb01862.x. PMID 2202752
- [Derived] McGarry A, Auinger P, Kieburtz KD, Bredlau AL, Hersch SM, Rosas HD. Suicidality Risk Factors Across the CARE-HD, 2CARE, and CREST-E Clinical Trials in Huntington Disease. Neurol Clin Pract. 2022 Apr;12(2):131-138. doi: 10.1212/CPJ.0000000000001161. PMID 35747889
- [Derived] McGarry A, McDermott MP, Kieburtz K, Fung WLA, McCusker E, Peng J, de Blieck EA, Cudkowicz M; Huntington Study Group 2CARE Investigators and Coordinators. Risk factors for suicidality in Huntington disease: An analysis of the 2CARE clinical trial. Neurology. 2019 Apr 2;92(14):e1643-e1651. doi: 10.1212/WNL.0000000000007244. Epub 2019 Mar 8. PMID 30850442
- [Derived] McGarry A, McDermott M, Kieburtz K, de Blieck EA, Beal F, Marder K, Ross C, Shoulson I, Gilbert P, Mallonee WM, Guttman M, Wojcieszek J, Kumar R, LeDoux MS, Jenkins M, Rosas HD, Nance M, Biglan K, Como P, Dubinsky RM, Shannon KM, O'Suilleabhain P, Chou K, Walker F, Martin W, Wheelock VL, McCusker E, Jankovic J, Singer C, Sanchez-Ramos J, Scott B, Suchowersky O, Factor SA, Higgins DS Jr, Molho E, Revilla F, Caviness JN, Friedman JH, Perlmutter JS, Feigin A, Anderson K, Rodriguez R, McFarland NR, Margolis RL, Farbman ES, Raymond LA, Suski V, Kostyk S, Colcher A, Seeberger L, Epping E, Esmail S, Diaz N, Fung WL, Diamond A, Frank S, Hanna P, Hermanowicz N, Dure LS, Cudkowicz M; Huntington Study Group 2CARE Investigators and Coordinators. A randomized, double-blind, placebo-controlled trial of coenzyme Q10 in Huntington disease. Neurology. 2017 Jan 10;88(2):152-159. doi: 10.1212/WNL.0000000000003478. Epub 2016 Dec 2. PMID 27913695

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Started | 303 | 306
Completed | 224 | 240
Not Completed | 79 | 66
Not completed — Death | 22 | 13
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 28 | 14
Not completed — Withdrawal by Subject | 18 | 29
Not completed — Physician Decision | 5 | 5
Not completed — Institutionalized | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo | Total
Number analyzed (Participants) | 303 | 306 | 609
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.9) | 50.7 (11.6) | 50.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 164 | 313
  Male | 154 | 142 | 296

OUTCOME MEASURES:

1. Primary Outcome: Joint Rank (Combination of Time to Death (for Subjects Who Died) and Change in Total Functional Capacity Score (TFC) From Baseline to Month 60 (for Subjects Who Survived))
Description: The primary outcome variable at the start of the trial was the change in TFC score from baseline to Month 60. The Data and Safety Monitoring Board recommended to the trial leadership that they reconsider how they accommodate missing data from subjects who die in their primary analysis of the change in TFC score. Based on these recommendations, the trial leadership changed the primary analysis to that of a joint rank approach. TFC consists of five ordinally scaled items assessing a person's capacity with: (1) occupation; (2) financial affairs; (3) domestic responsibilities; (4) activities of daily living; and (5) independent living. Total score ranges from zero (worst) to 13 (best).
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: rank
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
rank | 303.3 (173.1) | 306.7 (179.0)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; In this joint rank analysis, subjects are ranked from worst to best outcome with subjects who die being assigned the worst ranks (and ranked according to the time of death) and subjects who survive being ranked more favorably in the order of the change from baseline to Month 60 in TFC score; Test type: Superiority or Other; π hat = 0.494, 95% CI 2-sided [0.454 to 0.534] — π hat is the estimate of the probability π that a randomly selected subject treated with CoQ has a better outcome than a randomly selected subject treated with placebo. Under the null hypothesis of no effect of CoQ, π = 0.50

2. Secondary Outcome: Change in Total Functional Capacity (TFC) Score From Baseline to Month 60
Description: TFC consists of five ordinally scaled items assessing a person's capacity with: (1) occupation; (2) financial affairs; (3) domestic responsibilities; (4) activities of daily living; and (5) independent living. Total score ranges from zero (worst) to 13 (best).
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -4.53 (0.25) | -4.76 (0.24)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.23, 95% CI 2-sided [-0.44 to 0.91]

3. Secondary Outcome: Change in Functional Checklist Score From Baseline to Month 60
Description: The functional assessment checklist includes 25 questions about common daily tasks. A score of 1 is given for each "yes" reply and a score of 0 is given for each "no" reply (scale range is 0-25). Higher scores indicate better functioning.
Time Frame: Baseline and Month 60
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -7.93 (0.55) | -8.02 (0.54)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.09, 95% CI 2-sided [-1.40 to 1.58]

4. Secondary Outcome: Change in Independence Scale Score From Baseline to Month 60
Description: The independence scale assesses independence on a 0 to 100 scale with higher scores indicating better functioning.
Time Frame: Baseline and Month 60
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -26.30 (1.92) | -24.86 (1.90)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = -1.44, 95% CI 2-sided [-6.68 to 3.79]

5. Secondary Outcome: Change in Total Motor Score From Baseline to Month 60
Description: The motor section of the Unified Huntington's Disease Rating Scale (UHDRS) assesses motor features of Huntington disease with standardized ratings of oculomotor function, dysarthria, chorea, dystonia, gait, and postural stability. The total motor score is the sum of all the individual motor ratings, with higher scores (124) indicating more severe motor impairment than lower scores. The score ranges from 0 to 124.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | 18.06 (1.22) | 19.18 (1.18)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = -1.12, 95% CI 2-sided [-4.40 to 2.16]

6. Secondary Outcome: Change in Behavioral Frequency Score From Baseline to Month 60
Description: The Unified Huntington's Disease Rating Scale (UHDRS) behavioral subscale assesses frequency and severity of psychiatric-related symptoms, including depressed mood, apathy, low self-esteem/guilt, suicidal thoughts, anxiety, irritable behavior, aggressive behavior, obsessional thinking, compulsive behavior, delusions, and hallucinations. A total score was calculated by summing up all the individual behavioral frequency items (range 0-56) with higher scores representing more severe behavioral impairment.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | 1.39 (0.55) | 1.43 (0.53)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.04, 95% CI 2-sided [-1.48 to 1.39]

7. Secondary Outcome: Change in Behavioral Frequency x Severity Score From Baseline to Month 60
Description: The Unified Huntington's Disease Rating Scale (UHDRS) behavioral subscale assesses frequency and severity of psychiatric-related symptoms, including depressed mood, apathy, low self-esteem/guilt, suicidal thoughts, anxiety, irritable behavior, aggressive behavior, obsessional thinking, compulsive behavior, delusions, and hallucinations. The total score is the sum of the product of the individual behavioral frequency and severity items (range 0-176) with higher scores representing more severe behavioral impairment.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | 4.29 (1.52) | 5.06 (1.46)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.77, 95% CI 2-sided [-4.78 to 3.23]

8. Secondary Outcome: Change in Symbol Digit Modalities Test (SDMT) From Baseline to Month 60
Description: The SDMT assesses attention, visuoperceptual processing, working memory, and cognitive/psychomotor speed. The score is the number of correctly paired abstract symbols and specific numbers in 90 seconds with higher scores indicating better cognitive functioning.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -10.95 (0.66) | -11.36 (0.65)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = 0.41, 95% CI 2-sided [-1.32 to 2.14]

9. Secondary Outcome: Change in Verbal Fluency Test From Baseline to Month 60
Description: The verbal fluency test is typically considered a measure of executive function. The score is the number of correct words produced across three 1-minute trials.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -5.07 (0.79) | -4.47 (0.78)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = -0.60, 95% CI 2-sided [-2.71 to 1.51]

10. Secondary Outcome: Change in Stroop Interference Test - Color Naming From Baseline to Month 60
Description: Stroop Interference Test - color naming score is the total number of correct colors identified in 45 seconds and reflects processing speed.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -14.21 (1.00) | -14.51 (0.97)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-2.28 to 2.87]

11. Secondary Outcome: Change in Stroop Interference Test - Word Reading From Baseline to Month 60
Description: Stroop Interference Test - word reading score is the total number of correct words read in 45 seconds and reflects processing speed.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -15.25 (1.36) | -19.13 (1.32)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = 3.88, 95% CI 2-sided [0.31 to 7.44]

12. Secondary Outcome: Change in Stroop Interference Test - Interference From Baseline to Month 60
Description: Stroop Interference Test - interference score is the total number of correct items identified in 45 seconds and reflects an executive measure of inhibitory ability.
Time Frame: Baseline and Month 60
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
units on a scale | -7.57 (0.81) | -8.61 (0.79)
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Mean Difference (Net) = 1.04, 95% CI 2-sided [-1.10 to 3.18]

13. Secondary Outcome: Time to a Two-Point Decline in TFC Score or Death
Description: as for outcome 2
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: days to event
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
days to event | 553 [545 to 728] | 549 [395 to 726]
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.81 to 1.20]

14. Secondary Outcome: Time to a Three-Point Decline in TFC Score or Death
Description: as for outcome 2
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: days to event
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
days to event | 917 [760 to 1092] | 911 [737 to 1092]
Statistical Analysis 1: Comparison: A - Coenzyme Q10 2400 mg/Day vs B - Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.75 to 1.15]

15. Secondary Outcome: Number Completing Study at Assigned Dosage Level
Time Frame: 5 years
Measure: Number; unit: participants completing study on drug
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Number analyzed (Participants) | 303 | 306
participants completing study on drug | 98 | 108

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events were assessed at each visit by recording all voluntary complaints of the subject and by assessment of clinical features. Subjects were questioned regarding the occurrence of any adverse event since the last visit. All adverse events were recorded on an Adverse Event Log case report form.
Arm/Group | A - Coenzyme Q10 2400 mg/Day | B - Placebo
Serious Adverse Events (participants affected / at risk) | 76/303 | 83/306
Other Adverse Events (participants affected / at risk) | 276/303 | 280/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A - Coenzyme Q10 2400 mg/Day (N=303) | B - Placebo (N=306)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 3
HUNTINGTON'S DISEASE (Congenital, familial and genetic disorders) | 2 | 2
VERTIGO (Ear and labyrinth disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 2
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 2 | 0
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1
ABSCESS (Infections and infestations) | 1 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 2
GASTROENTERITIS (Infections and infestations) | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 2 | 5
SEPSIS (Infections and infestations) | 1 | 0
SKIN GRAFT INFECTION (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 0 | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 3 | 5
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
INJURY (Injury, poisoning and procedural complications) | 1 | 0
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 5
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
NOSE DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
CARCINOID TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
INFLAMMATORY CARCINOMA OF THE BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
CHOREA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 2
PARKINSONISM (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 3 | 2
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 | 0
AGGRESSION (Psychiatric disorders) | 2 | 2
AGITATION (Psychiatric disorders) | 1 | 1
ANXIETY (Psychiatric disorders) | 1 | 1
COMPLETED SUICIDE (Psychiatric disorders) | 4 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 1 | 0
DELUSION (Psychiatric disorders) | 1 | 2
DEPRESSION (Psychiatric disorders) | 2 | 6
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 | 1
MAJOR DEPRESSION (Psychiatric disorders) | 2 | 0
PANIC ATTACK (Psychiatric disorders) | 1 | 0
PARANOIA (Psychiatric disorders) | 1 | 0
PSYCHOTIC BEHAVIOUR (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 2 | 1
SUICIDAL BEHAVIOUR (Psychiatric disorders) | 1 | 1
SUICIDAL IDEATION (Psychiatric disorders) | 3 | 7
SUICIDE ATTEMPT (Psychiatric disorders) | 10 | 8
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 2
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
UPPER AIRWAY OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 0
DEEP BRAIN STIMULATION (Surgical and medical procedures) | 0 | 1
HAEMORRHOID OPERATION (Surgical and medical procedures) | 1 | 0
HERNIA REPAIR (Surgical and medical procedures) | 0 | 1
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 | 0
HYSTERECTOMY (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
SHOULDER ARTHROPLASTY (Surgical and medical procedures) | 1 | 0
SPINAL LAMINECTOMY (Surgical and medical procedures) | 1 | 0
SURGERY (Surgical and medical procedures) | 1 | 0
THYROIDECTOMY (Surgical and medical procedures) | 0 | 1
HYPOTENSION (Vascular disorders) | 2 | 0
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A - Coenzyme Q10 2400 mg/Day (N=303) | B - Placebo (N=306)
CONSTIPATION (Gastrointestinal disorders) | 26 | 22
DIARRHOEA (Gastrointestinal disorders) | 36 | 43
DYSPHAGIA (Gastrointestinal disorders) | 25 | 21
NAUSEA (Gastrointestinal disorders) | 31 | 24
VOMITING (Gastrointestinal disorders) | 25 | 23
FATIGUE (General disorders) | 19 | 16
BRONCHITIS (Infections and infestations) | 16 | 19
INFLUENZA (Infections and infestations) | 21 | 17
NASOPHARYNGITIS (Infections and infestations) | 27 | 34
SINUSITIS (Infections and infestations) | 14 | 19
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 23 | 27
URINARY TRACT INFECTION (Infections and infestations) | 33 | 46
CONTUSION (Injury, poisoning and procedural complications) | 10 | 21
FALL (Injury, poisoning and procedural complications) | 72 | 84
LACERATION (Injury, poisoning and procedural complications) | 14 | 23
WEIGHT DECREASED (Investigations) | 25 | 33
BALANCE DISORDER (Nervous system disorders) | 19 | 21
CHOREA (Nervous system disorders) | 37 | 44
DIZZINESS (Nervous system disorders) | 15 | 16
HEADACHE (Nervous system disorders) | 17 | 14
ANXIETY (Psychiatric disorders) | 36 | 42
DEPRESSION (Psychiatric disorders) | 61 | 66
INSOMNIA (Psychiatric disorders) | 35 | 64
IRRITABILITY (Psychiatric disorders) | 36 | 38
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 | 19

LIMITATIONS AND CAVEATS:
An interim analysis for futility revealed a conditional power of < 5% for the primary analysis, and the trial was halted in July, 2014. Only data collected prior to this time were included in the final analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No